CLINICAL TRIAL: NCT00734773
Title: A Pilot Study Incorporating Motexafin Gadolinium (MGd) Into High-dose Methotrexate (MTX)-Based Chemo-immunotherapy and Radiation for Patients With Newly Diagnosed Primary CNS Lymphoma
Brief Title: Pilot Study of MGd + High-dose MTX-Based Chemoimmunotherapy + RT for Newly Dx PCNSL
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Northwestern University (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Andrew M. Evens, Northwestern University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 05H7; STU00002443 (Other: Northwestern University IRB)
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Brain and Central Nervous System Tumors; Lymphoma; Neurotoxicity
Keywords: neurotoxicity; primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Lymphoma; Neurotoxicity Syndromes | interventions — Rituximab; Cytarabine; Methotrexate; motexafin gadolinium; Procarbazine; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Rituximab — Infusion will be given at week 2, week 4, week 6 and week 8. Infusions can be administered at an initial rate of 100 mg/hr, and increased by 100 mg/hr increments at 30-minute intervals, to a maximum of 400 mg/hr as tolerated.
  Other Names: Rituxan
Drug: Cytarabine — Administered by IV over 3 hours at a dose of 3 g/m2/day for 2 days given at week 17 and week 21.
  Other Names: Cytosar-U; Ara-c
Drug: Methotrexate — Administered by IV at dose of 3.5 grams/m2 on day 1 of week 1, week 3, week 5, week 7 and week 9; if CSF was positive it will also be given intrathecally on day 8 of week 1, week 3, week 5, week 7 and week 9.
  Other Names: MTX; Rheumatrex; Trexall
Drug: Motexafin gadolinium — * Administered to the first five patients enrolled on trial, MGd will be given at 5 mg/kg q day x2 doses (completed on 2 consecutive days 1 to 2 weeks prior to day of cycle 1) to be followed by a non-infused MRI (without contrast) 1-5 hours after 2nd MGd dose (to evaluate for MGd tumor selective uptake).
  * For induction chemotherapy, MGd 10 mg/kg will be given intravenously on day 8 of each cycle. MGd will be given immediately after Rituxan.
  * During radiation therapy, MGd will be administered at 5 mg/kg 2-5 hours prior to WBRT, daily for the first 10 days (fractions) and then every other day of radiation thereafter.
  Other Names: MGd
Drug: Procarbazine hydrochloride — Taken orally, 100 mg/m2 days 1-7 of the 1st, 3rd, and 5th cycles of induction therapy.
  Other Names: Matulane
Drug: Vincristine sulfate — Administered by IV at a dose of 1.4mg per meter squared on weeks 1, 3, 5, 7 and 9.
  Other Names: Vincasar PFS
Radiation: Radiation therapy — Given at weeks 11 through 16.
  Other Names: Whole Brain Radiation Therapy (WBRT)

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Radiation therapy uses high-energy x-rays to kill cancer cells. Motexafin gadolinium may make cancer cells more sensitive to radiation therapy and combination chemotherapy. Giving motexafin gadolinium together with chemotherapy, rituximab, and radiation therapy may kill more cancer cells.

PURPOSE: This phase II trial is studying the side effects of giving motexafin gadolinium together with combination chemotherapy, rituximab, and whole-brain radiation therapy and to see how well it works in treating patients with newly diagnosed primary central nervous system lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and efficacy of motexafin gadolinium (MGd) combined with high-dose methotrexate-based chemotherapy and radiotherapy in patients with newly diagnosed primary CNS lymphoma.
* Determine the toxicity of MGd and rituximab combined with high-dose methotrexate, procarbazine hydrochloride, and vincristine (MPV) in these patients.
* Determine the toxicity of MGd in combination with whole-brain radiotherapy (WBRT) in these patients.
* Determine the tumor-selective uptake of MGd.

Secondary

* Determine the overall response rate (complete remission [CR] and partial remission [PR]) in patients treated with pre-radiotherapy and chemo-immunotherapy (R-MPV with MGd).
* Determine the complete response rate in patients treated with this regimen.
* Determine the overall response rate (CR and PR) in patients who complete all MGd combined with high-dose methotrexate-based chemotherapy and WBRT.
* Determine the event-free and overall survival at 1 year of patients treated with this regimen.
* Determine the progression-free survival at 1 year of patients treated with this regimen.
* Evaluate the neurotoxicity of R-MVP with MGd based on pre- and post-treatment neuropsychologic testing.

OUTLINE:

* Tumor-selective imaging: Patients receive motexafin gadolinium (MGd) IV on days 1-2 beginning 1-2 weeks prior to induction therapy. They then undergo an MRI of the brain.
* Induction therapy: Patients receive methotrexate IV over 2-3 hours and vincristine IV on day 1 and rituximab IV over 5 hours and MGd IV over 30-60 minutes on day 8. Patients also receive oral procarbazine hydrochloride on days 1-7 of courses 1, 3, and 5. Treatment repeats every 14 days for 5 courses in the absence of disease progression or unacceptable toxicity. Patients with partial response receive an additional 2 courses of induction therapy.
* Chemoradiotherapy: Beginning 4 weeks after completion of induction therapy, patients undergo reduced-dose whole-brain radiotherapy for 6 weeks. Patients also receive MGd IV over 30-60 minutes, beginning 2-5 hours prior to radiotherapy, for 10 days and then every other day during radiotherapy.
* Consolidation therapy: After completion of chemoradiotherapy, patients receive cytarabine IV over 3 hours on days 1-2. Treatment repeats every 30 days for 2 courses.

After completion of study therapy, patients are followed every 3 months for the first year, every 3-4 months for the second year, every 4-6 months until the fifth year, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary CNS lymphoma (PCNSL) diagnosed by brain biopsy, CSF cytology, or vitreal biopsy

  * Newly diagnosed disease
  * Patients who have an inconclusive biopsy or who are not candidates for biopsy may be eligible provided they have a typical cranial MRI or CT scan (defined as the presence of hypo-, iso- or hyperdense parenchymal contrast-enhancing, usually homogeneously) mass lesion(s) and meet at least one of the following criteria:

    * Positive cerebrospinal fluid cytology for lymphoma or a monoclonal lymphocyte population as defined by cell surface markers
    * Biopsy of the vitreous or uvea demonstrating non-Hodgkin lymphoma
* Measurable (defined as reproducibly measurable disease in two perpendicular dimensions on radiologic study) or evaluable disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Life expectancy ≥ 8 weeks
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 2.0 mg
* SGOT ≤ 2 times upper limit of normal
* Serum creatinine ≤ 1.5 mg/dL OR creatinine clearance > 50 cc/min
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 6 months after completion of study therapy
* HIV negative
* No other active primary malignancy with the exception of basal cell carcinoma of the skin or cervical carcinoma in situ

PRIOR CONCURRENT THERAPY:

* No prior cranial irradiation
* No prior chemotherapy for CNS lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11

PRIMARY OUTCOMES:
Toxicity of motexafin gadolinium (MGd) and rituximab added to high-dose methotrexate, procarbazine hydrochloride, and vincristine (MPV) chemotherapy | Day 1 (every 2 weeks), After 5th cycle, After 7th cycle, Pre Radiation Theray, Post Radiation Therapy, and Post ara-c.
  To evaluate toxicity of motexafin gadolinium (MGd) and rituximab to high-dose methotrexate, procarbazine hydrochloride, and vincristine (MPV) chemotherapy at Day 1 (every 2 weeks), After 5th cycle, After 7th cycle, Pre Radiation Theray, Post Radiation Therapy, and Post ara-c.
Toxicity of MGd added to whole-brain radiotherapy (WBRT) | Day 1 (every 2 weeks), After 5th cycle, After 7th cycle, Pre Radiation Theray, Post Radiation Therapy, and Post ara-c.
  To evaluate the toxicity of MGd added to whole-brain radiotherapy (WBRT).
Tumor-selective uptake of MGd | Day 1 (every 2 weeks), After 5th cycle, After 7th cycle, Pre Radiation Theray, Post Radiation Therapy, and Post ara-c.
  To evaluate Tumor-selective uptake of MGd

SECONDARY OUTCOMES:
Overall response rate (complete remission [CR] and partial remission [CR]) to pre-radiation chemo-immunotherapy (R-MPV with MGd) | Every 3 months for the first year after completed treatment, every 4 months for the second year, every 6 months until the 5th year and then annually.
  MRI scan will be done with each neurologic evaluation. Neuropsychologic evaluation will be repeated approximately 6 months after the completion of therapy and at 6 months intervals thereafter for total of 2 years.
Complete response rate to pre-radiation chemo-immunotherapy (R-MPV with MGd) | Every 3 months after completion of treatment, exams every 3 months for the first year then every 4 - 6 months thereafter.
  Repeat CSF or ocular exam will be done 3 months after completion of treatment in those patients who had evidence of CSF or ocular involvement at diagnosis. CSF will be sampled at each visit. Ocular exams will occur every 3 months for the 1st year then every 4-6 months. Further exams will only be done as needed to rule out recurrent lymphoma.
Overall survival at 1 year | Every 3 months for the first year after completed treatment, every 4 months for the second year, every 6 months until the 5th year and then annually.
  To assess overall survival rate.
Event-free survival at 1 year | Every 3 months for the first year after completed treatment, every 4 months for the second year, every 6 months until the 5th year and then annually.
  To assess event-free survival rate.
Progression-free survival at 1 year | Every 3 months for the first year after completed treatment, every 4 months for the second year, every 6 months until the 5th year and then annually.
  To assess progression-free survival rate.
Neurotoxicity of R-MVP + MGd based on pre- and post-treatment neuropsychologic testing | At baseline
  MR perfusion and MR spectroscopy at baseline and serially when MRI imaging is done to assess response rates using these alternate forms of imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M. Evens, DO, MS, Principal Investigator — Robert H. Lurie Cancer Center; Jeffrey J. Raizer, MD, Principal Investigator — Robert H. Lurie Cancer Center